CLINICAL TRIAL: NCT01024036
Title: A Randomized, Double Blind, Placebo Controlled Study to Assess the Efficacy and Safety of CNTO 328 (Anti IL 6 Monoclonal Antibody) Plus Best Supportive Care Compared With Best Supportive Care in Subjects With Multicentric Castleman's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of CNTO328 Plus Best Supportive Care in Multicentric Castleman's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016705; CNTO328MCD2001 (Other: Janssen Research & Development, LLC); 2009-012380-34 (EudraCT Number)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-02

CONDITIONS: Multicentric Castleman's Disease
Keywords: Multicentric Castleman's Disease; MCD; CNTO 328; Best Supportive Care; Tumor; Symptomatic response; Pharmacokinetics; Interleukin-6; IL6
MeSH Terms: conditions — Multi-centric Castleman's Disease; Macular dystrophy, corneal type 1; Neoplasms | interventions — siltuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Siltuximab+best supportive care (BSC) (Experimental): Siltuximab 11 mg/kg will be administered as a 1-hour intravenous infusion every 3 weeks + BSC.
  Interventions: Drug: Siltuximab; Drug: Best Supportive Care (BSC)
- Placebo+BSC (Placebo Comparator): Placebo will be administered as a 1-hour intravenous infusion every 3 weeks + BSC. Participants who do not respond to placebo during the blinded treatment period will have option to crossover and receive siltuximab 11 mg/kg which will be administered by 1-hour intravenous infusion every 3 weeks + BSC during the unblinded treatment period.
  Interventions: Drug: Placebo; Drug: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Siltuximab — Siltuximab 11 mg/kg will be administered by 1-hour intravenous infusion every 3 weeks
  Other Names: CNTO 328
  Arms: Siltuximab+best supportive care (BSC)
Drug: Placebo — Placebo will be administered by 1-hour intravenous infusion every 3 weeks
  Arms: Placebo+BSC
Drug: Best Supportive Care (BSC) — BSC included treatment for effusions, antipyretics, antipuretics, antihistamines, pain medication, treatment for infections, transfusions, management of infusion-related reactions, and corticosteroids.

SUMMARY:
The purpose of this study is to demonstrate that CNTO 328 when administered in combination with best supportive care (BSC) is superior to BSC in terms of durable tumor and symptomatic response (complete response or partial response) among patients with Multicentric Castleman's Disease.

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), double blind (neither investigator nor the participant knows the treatment that the participant receives), placebo controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), study to assess the efficacy and safety of CNTO 328 plus BSC compared with BSC in patients with symptomatic Multicentric Castleman's Disease. The study mainly consists of 3 phases, including: the screening phase (majority of assessments performed within 28 days of first dose), the treatment phase (blinded and unblinded), and the follow up phase. In the blinded treatment phase, approximately 78 patients will be randomly assigned in 1:2 ratios to either of 2 treatment groups, ie, Placebo + BSC, or CNTO 328 + BSC. Participants receiving placebo + BSC during blinded treatment period who do not respond and have treatment failure will have the option to crossover and receive siltuximab + BSC during unbllinded treatent period. The follow up phase will be 3 months after last dose of study medication and the survival will be followed up until the study ends. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, patient-recorded temperature, and physical examination will be monitored throughout the study. The total study duration will be 5 years after the last patient starts study medication.

ELIGIBILITY:
Inclusion Criteria:

* Measurable and symptomatic Multicentric Castleman's Disease
* Adequate organ function as assessed by laboratory values evaluated by the investigator to determine eligibility prior to treatment
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Corticosteroids dose that does not exceed 1 mg/kg/day of prednisone, and has remained stable or decreased over the 4 weeks before treatment

Exclusion Criteria:

* Human Immunodeficiency Virus or Human Herpes Virus-8 positive
* Skin lesions as sole measurable manifestation of Multicentric Castleman's Disease
* Previous history of lymphoma
* Malignancies, except for adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or cancer other than lymphoma, from which the patient has been disease-free for 3 or more years
* Concurrent medical condition or disease that may interfere with study participation
* Prior exposure to Interleukin-6 or Interleukin-6 receptor targeted therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-03-18 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (56):
- United States (11):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Tampa, Florida
  - Boston, Massachusetts
  - Lansing, Michigan
  - Rochester, Minnesota
  - Chapel Hill, North Carolina
  - Greenville, South Carolina
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- East Melbourne, Australia
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (4):
  - Brasília
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Toronto, Canada
- China (5):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Shanghai
- Cairo, Egypt
- France (8):
  - Clermont-Ferrand
  - Grenoble
  - Lille
  - Montpellier
  - Paris
  - Rennes
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Berlin
  - Mainz
  - München
- Shatin, Hong Kong
- Budapest, Hungary
- India (2):
  - Hyderabad
  - Pune
- Israel (2):
  - Petah Tikva
  - Ramat Gan
- Pandan, Malaysia
- Rotterdam, Netherlands
- Auckland, New Zealand
- Oslo, Norway
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Seoul, South Korea
- Spain (2):
  - Barcelona
  - Madrid
- Taipei, Taiwan
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] van Rhee F, Rosenthal A, Kanhai K, Martin R, Nishimura K, Hoering A, Fajgenbaum DC. Siltuximab is associated with improved progression-free survival in idiopathic multicentric Castleman disease. Blood Adv. 2022 Aug 23;6(16):4773-4781. doi: 10.1182/bloodadvances.2022007112. PMID 35793409
- [Derived] Fajgenbaum DC, Uldrick TS, Bagg A, Frank D, Wu D, Srkalovic G, Simpson D, Liu AY, Menke D, Chandrakasan S, Lechowicz MJ, Wong RS, Pierson S, Paessler M, Rossi JF, Ide M, Ruth J, Croglio M, Suarez A, Krymskaya V, Chadburn A, Colleoni G, Nasta S, Jayanthan R, Nabel CS, Casper C, Dispenzieri A, Fossa A, Kelleher D, Kurzrock R, Voorhees P, Dogan A, Yoshizaki K, van Rhee F, Oksenhendler E, Jaffe ES, Elenitoba-Johnson KS, Lim MS. International, evidence-based consensus diagnostic criteria for HHV-8-negative/idiopathic multicentric Castleman disease. Blood. 2017 Mar 23;129(12):1646-1657. doi: 10.1182/blood-2016-10-746933. Epub 2017 Jan 13. PMID 28087540
- [Derived] van Rhee F, Wong RS, Munshi N, Rossi JF, Ke XY, Fossa A, Simpson D, Capra M, Liu T, Hsieh RK, Goh YT, Zhu J, Cho SG, Ren H, Cavet J, Bandekar R, Rothman M, Puchalski TA, Reddy M, van de Velde H, Vermeulen J, Casper C. Siltuximab for multicentric Castleman's disease: a randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2014 Aug;15(9):966-74. doi: 10.1016/S1470-2045(14)70319-5. Epub 2014 Jul 17. PMID 25042199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 79 participants were enrolled at 38 study centers in 19 countries. The first participant signed the informed consent on 09 Feb 2010, and the last participant's last visit for the primary analysis was 28 Feb 2013. The data until the end of study is presented here.
Pre-assignment Details: 79 participants were enrolled, randomized and treated during the blinded treatment period. 53 received siltuximab+best supportive care (BSC) and 26 received placebo+BSC.13 participants who did not respond to placebo+BSC during the blinded treatment period, received siltuximab+BSC during the unblinded treatment period.
Groups:
- Siltuximab + Best Supportive Care (BSC): Participants received siltuximab 11 milligram per kilogram (mg/kg) as a 1 hour intravenous (IV) infusion every 3 weeks along with BSC until treatment failure, discontinuation of treatment, withdrawal from study, or until 48 weeks after last participant started study treatment, whichever occurred earlier. Participants who discontinued treatment for any reason, completed End-of-Treatment (EOT) visit and entered Follow-up period. If a participant had documented treatment failure and wished to continue treatment, participant's treatment assignment was unblinded. Upon unblinding, if participant was assigned to siltuximab, study treatment was discontinued, and the participant completed EOT Visit and enter Follow up period (up to 3 months after last study drug intake) wherein participants were followed until death, lost to follow-up, withdrawal of consent, death of 50 percent (%) of participants, or end of the study, whichever occurred earlier.
- Placebo + Best Supportive Care (BSC): Participants received placebo as a 1-hour IV infusion every 3 weeks along with BSC until treatment failure, discontinuation of treatment, withdrawal from study, or until 48 weeks after last participant started study treatment, whichever occurred earlier. If a participant had documented treatment failure and wished to continue treatment, the participant's treatment assignment was unblinded. Upon unblinding placebo participants who received blinded treatment had an option to receive unblinded treatment with siltuximab. Participants who discontinued or completed treatment period up to Week 48 and who consented to enter follow-up period were continued to be followed up during the course of follow-up period (up to 3 months after last study drug intake) wherein participants were followed until death, lost to follow-up, withdrawal of consent, death of 50% of participants, or end of the study, whichever occurred earlier.
Period: Blinded Treatment
Arm/Group | Siltuximab + Best Supportive Care (BSC) | Placebo + Best Supportive Care (BSC)
Started | 53 | 26
Completed | 31 | 6
Not Completed | 22 | 20
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 16 | 14
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 4 | 3
Period: Unblinded Treatment
Arm/Group | Siltuximab + Best Supportive Care (BSC) | Placebo + Best Supportive Care (BSC)
Started | 0 (No participants in this group received treatment during unblinded treatment period) | 13 (Placebo participants had an option to receive siltuximab in unblinded treatment period)
Completed | 0 | 10
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Period: Follow-Up Period
Arm/Group | Siltuximab + Best Supportive Care (BSC) | Placebo + Best Supportive Care (BSC)
Started (Any participant who discontinued blinded/unblinded treatment could entered Follow-up period) | 14 | 6
Completed | 9 | 3
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 26 | 53 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.4) | 44.4 (13.32) | 45.5 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 23 | 27
  Male | 22 | 30 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 0 | 1 | 1
  BELGIUM | 0 | 3 | 3
  BRAZIL | 2 | 4 | 6
  CANADA | 1 | 0 | 1
  CHINA | 5 | 11 | 16
  EGYPT | 1 | 0 | 1
  FRANCE | 2 | 2 | 4
  GERMANY | 1 | 0 | 1
  HONG KONG | 2 | 3 | 5
  ISRAEL | 1 | 1 | 2
  NEW ZEALAND | 1 | 1 | 2
  NORWAY | 1 | 1 | 2
  RUSSIAN FEDERATION | 0 | 3 | 3
  SINGAPORE | 0 | 3 | 3
  SOUTH KOREA | 2 | 4 | 6
  SPAIN | 1 | 1 | 2
  TAIWAN | 1 | 3 | 4
  UNITED KINGDOM | 1 | 2 | 3
  UNITED STATES | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Durable Tumor and Symptomatic Response - by Independent Radiology Review
Description: Durable tumor and symptomatic response is complete response (CR) + partial response (PR). CR: complete disappearance of all measurable and evaluable disease (eg, pleural effusion) and resolution of baseline symptoms attributed to multicentric Castleman's disease, sustained for at least 18 weeks. PR: >=50 percent decrease in sum of the product of the diameters of indicator lesion(s), with at least stable disease in all other evaluable disease in the absence of treatment failure sustained for at least 18 weeks. The statistical analysis shows difference in symptomatic response rate (siltuximab+best supportive care [BSC] minus Placebo+BSC).
Time Frame: From Day 1 of Cycle 1 of treatment with study medication until treatment failure or discontinuation of treatment or withdrawal from study, or up to 48 weeks after last participant started study medication(approximately 3 years), whichever occurred earlier
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Percentage of participants | 0 | 34
Statistical Analysis 1: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Null hypothesis: there is no difference in the durable tumor and symptomatic response rate between the 2 treatment arms; Test type: Superiority or Other; p = 0.0012, Cochran-Mantel-Haenszel; Adjusted for the stratification factor: corticosteroid use; difference in the response rate = 34, 95% CI 2-sided [11.1 to 54.8]
Statistical Analysis 2: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Null hypothesis: there is no difference in the durable tumor and symptomatic response rate between the 2 treatment arms; Test type: Superiority or Other; p = 0.0004, Fisher Exact; Without adjusting for the stratification factor: corticosteroid use; difference in the response rate = 34.0, 95% CI 2-sided [11.1 to 54.8]

2. Secondary Outcome: Median Duration of Tumor and Symptomatic Response - by Independent Radiology Review
Description: Duration of tumor and symptomatic response is defined as time from first documentation of tumor and symptomatic response (CR or PR) to treatment failure. Whenever possible, treatment failure documented by the appearance of new lesions should be confirmed by histologic examination of the new lesions. Symptomatic response is complete response (CR) + partial response (PR). CR: complete disappearance of all measurable and evaluable disease (eg, pleural effusion) and resolution of baseline symptoms attributed to multicentric Castleman's disease, sustained for at least 18 weeks. PR: >=50 percent decrease in sum of the product of the diameters of indicator lesion(s), with at least stable disease in all other evaluable disease in the absence of treatment failure sustained for at least 18 weeks.
Time Frame: From the date when durable tumour and symptomatic response is achieved until treatment failure, as assessed until 48 weeks after the last participant started study treatment (approximately 3 years)
Population: All randomized participants who achieved durable tumor and symptomatic response during blinded treatment period as per independent review.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 0 | 18
Days |  | 383.0 [232 to 676]

3. Secondary Outcome: Percentage of Participants Who Achieved Complete Response (CR) + Partial Response (PR) (Tumor Response Rate) - by Independent Radiology Review
Description: Overall tumor response is CR + PR assessed according to Cheson criteria. CR: complete disappearance of all measurable and evaluable disease (eg, pleural effusion). PR: a >=50 percent decrease in sum of the product of the diameters of index lesion(s), with at least stable disease in all other evaluable disease. Statistical analysis shows difference of overall response rates (siltuximab+best supportive care [BSC] minus Placebo+BSC).
Time Frame: From Day 1 of Cycle 1 until the date when durable tumour and symptomatic response is achieved, as assessed up to 48 weeks after the last participant started study treatment (approximately 3 years)
Population: Response-evaluable Population: included participants who received at least 1 administration of siltuximab/placebo and had at least 1 post-baseline radiologic disease evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Percentage of participants | 3.8 | 37.7
Statistical Analysis 1: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel; Difference in overall response rates = 33.9, 95% CI 2-sided [11.1 to 54.8]

4. Secondary Outcome: Median Duration of Tumor Response - by Independent Radiology Review
Description: Duration of tumor response is defined as time from first documentation of tumor response to tumor progression. Tumour response is complete response (CR) + partial response (PR) as assessed according to Cheson criteria. CR: complete disappearance of all measurable and evaluable disease (eg, pleural effusion). PR: a >=50 percent decrease in sum of the product of the diameters of index lesion(s), with at least stable disease in all other evaluable disease. Statistical analysis shows difference of overall response rates (siltuximab+best supportive care [BSC] minus Placebo+BSC).
Time Frame: From the date when tumour response is achieved until tumour progression, as assessed up to 48 weeks after the last participant started study treatment (approximately 3 years)
Population: All randomized participants who achieved tumor response during blinded treatment period as per independent review.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 1 | 20
Days | 70 [70 to 70] | 356 [55 to 674]

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from randomization until the participant fails treatment. Treatment failure was defined as any of the following: a sustained increase from baseline in disease related symptoms >=Grade 2 persisting for at least 3 weeks despite best supportive care (BSC); onset of any new disease related Grade 3 or higher symptom despite BSC; sustained (ie, at least 3 weeks) deterioration in performance status (increase from baseline in Eastern Cooperative Oncology Group Performance Status by more than 1 point) despite BSC; radiologic progression, as measured by modified Cheson criteria; Initiation of any other therapy intended to treat multicentric Castleman's disease ie, prohibited treatments. Statistical analysis shows difference in treatment failure rate (siltuximab+BSC minus Placebo+BSC).
Time Frame: From the date of randomization until a participant fails treatment, as assessed up to 48 weeks after the last participant started study treatment (approximately 3 years), whichever occurred earlier
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Days | 134 [85 to NA] — The upper limit was not estimable due to insufficient number of participants with event. | NA [378 to NA] — Median time to treatment failure was not estimable due to insufficient number of participants with event.
Statistical Analysis 1: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0084, Log Rank; Hazard Ratio (HR) = 0.418, 95% CI 2-sided [0.214 to 0.815] — Hazard ratio and 95% CI from a Cox proportional hazards model

6. Secondary Outcome: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 15 Gram Per Liter (g/L) Hemoglobin at Week 13 (Hemoglobin Response Rate)
Description: Hemoglobin response rate is defined as percentage of participants who achieved >= 15 g/L hemoglobin at Week 13.
Time Frame: Week 13
Population: Hemoglobin response-evaluable population: participants who received at least 1 siltuximab/placebo administration and have a baseline hemoglobin that is below the lower limit of normal as per local laboratory specifications (within 2 weeks before starting treatment) and at least 1 postbaseline hemoglobin evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 11 | 31
Percentage of participants | 0 | 61.3
Statistical Analysis 1: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Difference of hemoglobin response rates = 61.3, 95% CI 2-sided [28.3 to 85.1] — Difference in hemoglobin response rates is equal to hemoglobin response rate for siltuximab+best supportive care [BSC] arm minus hemoglobin response rate for Placebo+BSC arm

7. Secondary Outcome: Percentage of Participants Who Achieved >= 20 g/L Hemoglobin at Week 13 (Hemoglobin Response Rate)
Description: Hemoglobin response rate is defined as percentage of participants who achieved >= 20 g/L hemoglobin at Week 13.
Time Frame: Week 13
Population: Hemoglobin response-evaluable population: participants who received at least 1 siltuximab/placebo administration and have a baseline hemoglobin that is below the lower limit of normal as per local laboratory specifications (within 2 weeks before starting treatment) and at least 1 post-baseline hemoglobin evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 11 | 31
Percentage of participants | 0 | 41.9
Statistical Analysis 1: Comparison: Placebo + Best Supportive Care (BSC) vs Siltuximab + Best Supportive Care (BSC); Test type: Superiority or Other; p = 0.0195, Cochran-Mantel-Haenszel; Difference of hemoglobin response rates = 41.9, 95% CI 2-sided [7.8 to 70.7] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Participants Who Discontinued Corticosteroids
Description: Percentage of participants who discontinued corticosteroids during blinded treatment period and who were dependent on corticosteroids at baseline (Day 1 of Cycle 1).
Time Frame: From Day 1 of Cycle 1 until 48 weeks after the after the last participant started study treatment (approximately 3 years)
Population: All randomized participants who were dependent on corticosteroids at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 9 | 13
Percentage of participants | 11.1 | 30.8

9. Secondary Outcome: 6-year Survival Rate
Description: Overall survival was defined as percent chance of survival of participants who were still alive at 6 years from time of first study treatment was analyzed.
Time Frame: until 6 years
Population: Safety Analysis set included all randomized participants who received at least 1 dose of study agent.
Measure: Median (95% Confidence Interval); unit: Percent chance of survival
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Percent chance of survival | 79.5 [57.5 to 91.0] | 86.3 [71.9 to 93.6]

10. Secondary Outcome: Median Time Required to Achieve >=1 Point Decrease in the Multicentric Castleman's Disease Symptom Scale (MCD-SS) Score From Baseline
Description: A patient-reported symptom scale. Symptom presence/absence and severity are noted on an anchor-based numeric scale. Scores range from 1 (very mild) to 5 (very severe).
Time Frame: From Day 1 of Cycle 1 (baseline) until 48 weeks after the last participant started study treatment (approximately 3 years)
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Days | 262 [40 to NA] — The upper limit was not estimable due to insufficient number of participants with event. | 85 [22 to 379]

11. Secondary Outcome: Median Time Required to Achieve >=3-point Increase in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scores From Baseline
Description: The FACIT-F, a 13-item instrument, was designed to measure patient-reported fatigue. It is one of the suite of FACIT instruments developed for outcomes in cancer. Concepts measured in the scale include tiredness, weakness, and difficulty conducting usual functional activities or social interaction due to fatigue. Response options range from "not at all" (0) to "very much" (4), and yield a summary score. Total FACIT-F score is the sum of 13 items, ranging from 0 (not at all) to 52 (very much). Higher scores represent better outcomes.
Time Frame: as for outcome 10
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Days | 22 [8 to 64] | 15 [8 to 23]

12. Secondary Outcome: Median Time Required to Achieve >=5-point Increase in the Short-Form-36 (SF-36) Physical Component Summary (PCS) Scores From Baseline
Description: SF-36 is a questionnaire and PCS is a part of subscale assessing physical functioning, role-physical, bodily pain, and general health. The scores range from 0 (worst score) to 100 (best score), with a higher score indicating better quality of life.
Time Frame: as for outcome 10
Population: Intent-to-treat (ITT) population: all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Best Supportive Care (BSC) | Siltuximab + Best Supportive Care (BSC)
Number analyzed (Participants) | 26 | 53
Days | NA [169 to NA] — Median time was not estimable due to insufficient number of participants with event. | 420 [106 to NA] — The upper limit was not estimable due to insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Safety Analysis set included all participants who received at least 1 dose of study drug in blinded and unblinded treatment period until 48 weeks after the last subject started study treatment (approximately 3 years). Participants who continued in the study from Week 48 through the end-of-study (5 years after the last participant started study treatment) were included in the Follow-up analysis set.
Groups:
- Placebo + Best Supportive Care (BSC) (Blinded): Participants received placebo as a 1-hour intravenous infusion every 3 weeks along with BSC until treatment failure, discontinuation of treatment, withdrawal from the study, or until 48 weeks after the last participant started study treatment, whichever occurred earlier. Participants who discontinued or completed treatment period up to Week 48, and who consented to enter the follow-up period were continued to be followed up during the course of follow-up period.
- Siltuximab + Best Supportive Care (BSC) (Blinded): Participants received siltuximab 11mg/kg as a 1-hour intravenous infusion every 3 weeks along with BSC until treatment failure, discontinuation of treatment, withdrawal from the study, or until 48 weeks after the last participant started study treatment, whichever occurred earlier. Participants who discontinued treatment for any reason completed the end-of-treatment visit and entered the follow-up period.
- Siltuximab + Best Supportive Care (BSC) (Unblinded): Participants who had documented treatment failure and wished to continue treatment, their treatment assignment was unblinded. Upon unblinding placebo participants who received blinded treatment had an option to receive unblinded treatment with siltuximab during the unblinded treatment period.
- Placebo + BSC (Follow-up Period): No study treatment was administered during the follow-up period (up to 3 months after last study agent administration [placebo as a 1 hour IV infusion every 3 weeks along with BSC]) and participants were followed until death, lost to follow up, withdrawal of consent, death of 50 % of participants, or the end of the study, whichever occurred earlier.
- Siltuximab + BSC (Follow-up Period): No study treatment was administered during the follow-up period (up to 3 months after last study agent administration [siltuximab 11mg/kg as a 1 hour IV infusion every 3 weeks along with ]) and participants were followed until death, lost to follow up, withdrawal of consent, death of 50 % of participants, or the end of the study, whichever occurred earlier.
Arm/Group | Placebo + Best Supportive Care (BSC) (Blinded) | Siltuximab + Best Supportive Care (BSC) (Blinded) | Siltuximab + Best Supportive Care (BSC) (Unblinded) | Placebo + BSC (Follow-up Period) | Siltuximab + BSC (Follow-up Period)
Serious Adverse Events (participants affected / at risk) | 7/26 | 12/53 | 4/13 | 1/6 | 3/14
Other Adverse Events (participants affected / at risk) | 25/26 | 53/53 | 13/13 | 5/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Best Supportive Care (BSC) (Blinded) (N=26) | Siltuximab + Best Supportive Care (BSC) (Blinded) (N=53) | Siltuximab + Best Supportive Care (BSC) (Unblinded) (N=13) | Placebo + BSC (Follow-up Period) (N=6) | Siltuximab + BSC (Follow-up Period) (N=14)
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Mycobacterium Test (Investigations) | 1 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Poems Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureteral Disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1 | 0
Pain Management (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Best Supportive Care (BSC) (Blinded) (N=26) | Siltuximab + Best Supportive Care (BSC) (Blinded) (N=53) | Siltuximab + Best Supportive Care (BSC) (Unblinded) (N=13) | Placebo + BSC (Follow-up Period) (N=6) | Siltuximab + BSC (Follow-up Period) (N=14)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 4 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 2 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 8 | 1 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 2 | 0 | 0
Noninfective Conjunctivitis (Eye disorders) | 2 | 1 | 1 | 1 | 0
Periorbital Oedema (Eye disorders) | 2 | 3 | 2 | 0 | 1
Vision Blurred (Eye disorders) | 1 | 3 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 4 | 1 | 0 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 8 | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 5 | 1 | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 6 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 13 | 4 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 5 | 3 | 1 | 0
Tongue Ulceration (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 3 | 0 | 2
Chest Pain (General disorders) | 2 | 0 | 1 | 0 | 0
Face Oedema (General disorders) | 1 | 6 | 1 | 1 | 1
Fatigue (General disorders) | 14 | 18 | 8 | 2 | 4
Generalised Oedema (General disorders) | 4 | 7 | 2 | 2 | 1
Localised Oedema (General disorders) | 3 | 11 | 2 | 2 | 1
Malaise (General disorders) | 7 | 15 | 6 | 2 | 5
Oedema Peripheral (General disorders) | 8 | 19 | 4 | 3 | 5
Pain (General disorders) | 2 | 3 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 6 | 2 | 0 | 3
Hepatic Function Abnormal (Hepatobiliary disorders) | 3 | 2 | 3 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 4 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 9 | 1 | 1 | 2
Rash Pustular (Infections and infestations) | 2 | 4 | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 20 | 4 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0
Blood Albumin Decreased (Investigations) | 3 | 1 | 2 | 1 | 1
Serum Ferritin Decreased (Investigations) | 0 | 3 | 0 | 0 | 0
Weight Decreased (Investigations) | 7 | 4 | 3 | 3 | 2
Weight Increased (Investigations) | 0 | 11 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 9 | 4 | 3 | 4
Enzyme Abnormality (Metabolism and nutrition disorders) | 4 | 1 | 4 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 7 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 7 | 1 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 6 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 6 | 0 | 0 | 2
Peripheral Motor Neuropathy (Nervous system disorders) | 4 | 6 | 2 | 2 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 13 | 5 | 3 | 3
Insomnia (Psychiatric disorders) | 2 | 5 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 2 | 2 | 1 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 2 | 4 | 2 | 1 | 2
Oedema Genital (Reproductive system and breast disorders) | 2 | 3 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 4 | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2 | 3 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 10 | 5 | 2 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 9 | 4 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 22 | 4 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 18 | 3 | 2 | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 1
Flushing (Vascular disorders) | 2 | 2 | 2 | 0 | 0
Hypertension (Vascular disorders) | 3 | 4 | 3 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Idiopathic Orbital Inflammation (Eye disorders) | 1 | 0 | 1 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 2 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Tongue Coated (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 1 | 0 | 0
Infusion Site Extravasation (General disorders) | 1 | 0 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Oral Candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood Folate Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood Iron Decreased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood Phosphorus Increased (Investigations) | 0 | 1 | 0 | 0 | 1
Haemoglobin Increased (Investigations) | 0 | 2 | 0 | 0 | 1
Iron Binding Capacity Total Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Iron Binding Capacity Unsaturated Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Platelet Count Increased (Investigations) | 1 | 0 | 0 | 1 | 0
Protein Total Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Protein Total Increased (Investigations) | 1 | 0 | 1 | 1 | 0
Protein Urine Present (Investigations) | 1 | 0 | 0 | 1 | 0
Reticulocyte Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Reticulocyte Percentage Decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Vitamin B12 Decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Scrotal Swelling (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days